CLINICAL TRIAL: NCT01948336
Title: Phase 4 THE EFFECTS OF DEXMEDETOMIDINE ON EARLY STAGE RENAL FUNCTIONS IN PEDIATRIC PATIENTS UNDERGOING CARDIAC ANGIOGRAPHY USING NON- IONIC CONTRAST MEDIA: A DOUBLE- BLIND, RANDOMIZED CLINICAL TRIAL
Brief Title: The Effects of Dexmedetomidine on Early Stage Renal Functions in Pediatric Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Adnan Bayram, Assisstant Professor, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2011-200
Record Dates: First submitted 2013-09-14; First posted 2013-09-23 (Estimated); Last update posted 2013-09-23 (Estimated); Status verified 2013-09

CONDITIONS: Renal Function Disorder; Hemodynamic Instability
Keywords: Contrast-induced nephropathy, Dexmedetomidine, Endothelin-1
MeSH Terms: interventions — Dexmedetomidine; Ketamine; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): The patients in group C (control) (n=30) were bolused with 1 mg kg-1 ketamine (Ketalar®, Eczacibasi, Luleburgaz, Turkey) (IV) and 1 mg kg-1 propofol (Propofol 1% Fresenius, Fresenius Kabi Deutschland, Bad Homburg, Germany) (IV) followed by 1 mg kg-1 hour-1 ketamine (IV) and 50 µg kg-1 min-1 propofol (IV) infusion. Additionally a loading dose of 1 ml kg-1 D5 0.3% NaCl IV given over 10 minutes, followed by 0.5 ml kg-1 hour-1 IV D5 0.3% NaCl infusion were administered.
  Interventions: Drug: Ketamine; Drug: Propofol
- Dexmedetomidine (Active Comparator): The patients in group D (dexmedetomidine) (n=30) were bolused with 1mg kg-1 ketamine (IV), 1mg kg-1 propofol (IV) followed by 1 mg kg-1 hour-1 ketamine (IV) and 50 µg kg-1 min-1 propofol (IV) infusion. Additionally a loading dose of 1 µg kg-1 dexmedetomidine (Precedex Abbott Labs, North Chicago, IL) IV given over 10 minutes, followed by 0.5 µg kg-1 hour-1 IV dexmedetomidine infusion were administered. Dexmedetomidine was prepared as a 1 µg ml-1 solution using D5 0.3% NaCl solution.
  Interventions: Drug: Dexmedetomidine; Drug: Ketamine; Drug: Propofol

INTERVENTIONS:
Drug: Dexmedetomidine — a loading dose of 1 µg kg-1 dexmedetomidine (Precedex Abbott Labs, North Chicago, IL) IV given over 10 minutes, followed by 0.5 µg kg-1 hour-1 IV dexmedetomidine infusion were administered. Dexmedetomidine was prepared as a 1 µg ml-1 solution using D5 0.3% NaCl solution.
  Other Names: Precedex
  Arms: Dexmedetomidine
Drug: Ketamine — ketamine was bolused with 1 mg kg-1(IV) and followed by 1 mg kg-1 hour-1 ketamine IV infusion during the procedure.
  Other Names: Ketalar
Drug: Propofol — propofol was bolused 1 mg kg-1 and 50 µg kg-1 min-1 propofol (IV) infusion during the procedure.
  Other Names: Pofol

SUMMARY:
The aim of this study is to evaluate the effect of dexmedetomidine infusion on early stage renal function.

DETAILED DESCRIPTION:
Background: Contrast-induced nephropathy is the third most common cause of acute renal failure in hospitalized patients in all age groups. In this study we aimed to investigate the effects of dexmedetomidine on early stage renal function in pediatric patients undergoing cardiac angiography.

Methods: 60 pediatric patients between 6 and 72 months of age undergoing cardiac angiography were included in the study. Patients were divided into two groups. The patients in both groups were administered 1mgkg-1 ketamine, 1mgkg-1 propofol as bolus and followed by 1 mgkg-1hour-1 ketamine and 50 µgkg-1min-1 propofol infusion. Additionally, a loading dose of 1 µgkg-1 dexmedetomidine given over 10 minutes followed by 0.5 µgkg-1hour-1 dexmedetomidine infusion to patients in group D. The patients were evaluated for NGAL, creatinine, renin, endothelin-1, TAS and TOS blood levels before the procedure and 6th and 24th hours after the procedure. pRIFLE criteria were used to define CIN and its incidence in the study.

ELIGIBILITY:
Inclusion Criteria:

* 6 and 72 months children
* scheduled for cardiac angiography

Exclusion Criteria:

* patients with renal failure or diabetes mellitus, patients who were on nephrotoxic and vasoactive drugs simultaneously, patients with decompensated congestive heart failure and patients who had been administered contrast media in the last two weeks

Ages: 6 Months to 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2012-04; Primary Completion 2013-04 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Renal Functions, | Baseline, changes from baseline at 6th and 24th hours after the cardiac angiography
  The patients were evaluated for complete blood count and blood levels of creatinine (Cr), Neutrophil Gelatinase-Associated Lipocalin (NGAL), renin, endothelin-1, total antioxidant status (TAS) and total oxidant status (TOS) before the procedure and 6 and 24 hours after the procedure.

SECONDARY OUTCOMES:
Blood Pressure | Up to 24 hours
  After the patients were taken to the pediatric cardiac catheterization laboratory, mean arterial pressure (MAP), heart rate (HR), peripheral oxygen saturation (SpO2).
Heart rate | Up to 24 hours
  After the patients were taken to the pediatric cardiac catheterization laboratory, mean arterial pressure (MAP), heart rate (HR), peripheral oxygen saturation (SpO2).
peripheral oxygen saturation | Up to 24 hours
  After the patients were taken to the pediatric cardiac catheterization laboratory, mean arterial pressure (MAP), heart rate (HR), peripheral oxygen saturation (SpO2).

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Bayram, Asst. Prof., Study Chair — TC Erciyes University